CLINICAL TRIAL: NCT01760356
Title: Study of Pharmacodynamic, Pharmacokinetic and Pharmacogenetic Relationships of Anticalcineurin Drugs: Tacrolimus and Cyclosporin in Liver Transplant Recipients.
Brief Title: Study of PD/PK/PG Relationships of Tacrolimus and Cyclosporin in Liver Transplant Patients
Acronym: 3PIGREF
Status: Terminated | Type: Observational
Sponsor: UDA Centro Nacional Hepato-Bilio-Pancreático (Other)
Collaborators: INSERM UMR-S850, Limoges, France (Unknown); University Hospital, Limoges (Other); PEDECIBA, Uruguay (Unknown); Universidad de la Republica (Other); ANII (Agencia Nacional de Investigación e Innovación), Uruguay (Unknown); Scientific Cooperation Service, French Embassy, Uruguay (Unknown); Hospital Central de las Fuerzas Armadas, Uruguay (Unknown); ECOS Sud Program France-Uruguay (Unknown); National Center for Liver Transplantation, Uruguay (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3PIGREF- 2009 -1165
Record Dates: First submitted 2012-12-01; First posted 2013-01-04 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: End Stage Liver Disease; Rejection; Infection; Malignancy; Toxicity; Diabetes
Keywords: Liver transplantation; Calcineurin inhibitors; Pharmacodynamic biomarkers; Calcineurin pathway; Tacrolimus; interindividual variability
MeSH Terms: conditions — End Stage Liver Disease; Rejection, Psychology; Infections; Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Samples from whole blood: PBMC,DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy Volunteers No treatment: This is set as reference a cohort of untreated healthy volunteers, over which will be measured the biomarkers to determine the baseline. Implies PBMC ex-vivo exposure to Tacrolimus prior all cell incubations to study ex-vivo PD in stimulated conditions with mitogens to identify potential genetic sources of interindividual variability in physiological conditions Number proposed 30.
- Liver Transplant Patients on Tacrolimus: To explore PD/PG/PK relationships of TAC residual PD activities ex-vivo in stimulated and non-stimulated conditions in liver recipients.
  The number proposed is 50.
- Waiting List for Liver Transplantation: To study the ex-vivo PD response to TAC in stimulated and non-stimulated conditions and the potential genetic sources of PD variability in pathological conditions.
  The number proposed is 12.
- Liver Transplant Patients on Cyclosporine: To explore PD/PG/PK relationships of CsA residual PD activities ex-vivo in stimulated and non-stimulated conditions in liver recipients.
  The number proposed is 10.
- Longitudinal Cohort: Patients form the waiting list for liver transplantation will be enrolled and monitored at different times after transplantation to study the relationships between TAC PD and the clinical responses.
  The number proposed is 20.

SUMMARY:
To search for suitable pharmacodynamic biomarkers, i.e., with high specificity for calcineurin inhibition and most affected by inter-individual variability, our works aimed at exploring the pharmacodynamics of CNI, the strength and variability of signal translation along the calcineurin pathway, as well as the steps where sources of internal (genetic) or external variability are the most influential.

In order to achieve this, we assessed simultaneously NFAT1 translocation into the nucleus of peripheral blood mononuclear cells (PBMC) (NFTA1 being the main NAFT isoform in resting and activated lymphocytes), the intracellular expression of IL-2 in CD3+, CD4+ and CD8+ T cell subsets and the membrane expression of CD25 (IL-2Rα), a surface marker of T cells activation, in T cells at large. A non-interventional clinical trial was set up in healthy volunteers, patients registered on a liver transplantation waiting list (WLP) and liver transplant recipients (LTR). A different question was addressed in each group: The healthy volunteer study (n=35): explored TAC PD along the calcineurin pathway by exposing PBMC ex-vivo; modelled signal translation along this cascade; examined the interindividual variability of TAC PD parameters; and investigated the sources of the variability observed and their contribution at each step of the calcineurin pathway. Furthermore, it allowed us to evaluate the analytical variability of our techniques as well as the intra-individual variability of TAC PD parameters. WLP (n=19) were enrolled to confirm in patients with liver diseases the results obtained in healthy volunteers, as well as to test the potential influence of their initial disease on the ex-vivo pharmacodynamics of TAC. The aims of the transversal study of LTR on CNI (n=80) were to further explore the interindividual variability in the PD of CNI in realistic clinical conditions, i.e. in situations of residual PD activities under tacrolimus or cyclosporine exposure, and the potential pharmacogenetic (PG) sources of such variability. The (still small) group of liver transplant patients (n=9) enrolled immediately before transplantation and followed-up with serial monitoring along the first year post-transplantation was intended to explore the relationships between CNI PD and clinical responses.

DETAILED DESCRIPTION:
The research will be conducted under the rules of Good Clinical Practice, Good Laboratory Practice of the International Conference on Harmonisation (ICH)and the Principles of Declaration of Helsinki.

Groups of study are included once inclusion/exclusion criteria were verified and after written informed consent was given: healthy volunteers, patients of the waiting list for liver transplantation, liver transplant recipients on tacrolimus and cyclosporine and a longitudinal cohort of patients enrolled since the waiting list for transplantation.

From this instance proceed the sampling plan. Considering potential dropouts or withdrawals during the study, the intention is to recruit an additional 10% to compensate for the cohorts, as they allow.

The study design does not suppose applying masking methods, since it is an open study.

All data required in the registration forms will be recorded, however in case of persistent failure, will be properly documented the reasons for the absence. Each instance will merit a particular analysis, dated and signed.

Models could be used to estimate the impact of bias due to potential missing data, and if applicable will be complemented with a sensibility analysis.

Loading data will be conducted electronically. Data will be validated according to the data management plan, jointly defined by the principal investigator and the biostatistician, including freezing and thawing processes.

Pharmacokinetic, pharmacogenetic and pharmacodynamic modeling will be done using R software.

Data back ups will be run everyday, and will be archived on tape and a USB storage drive.

Besides self monitoring procedures, the study may be audited by the health authority (during the course of the study or even when it is completed), to assess compliance with the standards of Good Clinical Practice.

Atypical results if any, will be handled according to the criteria of results outside of specification. If re-analysis of samples will occur, they will be properly documented.

Sample size calculation includes the percentage of occurrence of acute cellular rejection and adverse events, as reported by the National Liver Transplant Program and the possible rates of abandonment or premature retirement of the in study subjects.

Under national rates, will be studied at least 30 healthy volunteers, 50 patients and 12 patients with end stage liver disease enlisted for liver transplantation, with serial follow-up during the first year.

Statistical analysis will be performed according to the principle of "intention to treat", and will be the responsible for at least one specialist in biostatistics.

It will be developed a descriptive analysis of all variables collected. Categorical variables will be expressed in percentages and number of observations. Continuous variables will be expressed as mean and coefficient of variation or median and 25th and 75th percentiles, minimum and maximum. Lof transformations will be held whenever needed.

The variables will be compared between groups according to the patient's original listing (intention to treat). They will be calculated and presented the estimated relative risks and their effect with 95% confidence intervals.

For comparison of categorical variables, it will be used the Chi-square test or Fisher's exact test as appropriate.

For comparison of continuous variables, it will be used the test "t" of Student.

For variables that develop with time, they will be represented by Kaplan-Meier curves and compared using the "log-rank" test. Their relative risk with 95% confidence interval will be calculated.

To identify variables associated with different responses multivariate linear analysis, logistic or Cox proportional will be used.

All analyzes will be performed with hypothesis testing and a 2-tailed significance level of 5%.

The program used will be R. Multivariate analysis will be held corrected according Bonferroni's criteria.

We have established standard operating procedures to describe blood collection instances, biological fluids sampling circuit, evaluation of the candidates to include in the study, verification of the inclusion criteria, monitoring of patients during the study, record of undesirable events and report of adverse drug reactions, terminating tracking.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Age: 18 to 70 years.
* Ethnicity: Hispanic, African American.
* Gender: male and female.
* Condition: healthy.
* Informed consent: granted and signed informed consent at the time of inclusion and agreement to comply with all the procedures included in the protocol.

Waiting List Patients:

* Age: 18 to 70 years.
* Ethnicity: Hispanic, African American.
* Gender: male and female.
* Being active on the waiting list for liver transplantation
* Informed consent: granted and signed at the time of inclusion and agreement to comply with all the procedures included in the protocol.

Transplant Patients:

* Age: 18 to 70 years.
* Ethnicity: Hispanic, African American.
* Gender: male and female.
* Drug therapy: cyclosporine or tacrolimus, with or without mycophenolic acid derivatives and/or corticosteroids.
* Informed consent: granted and signed at the time of inclusion and agreement to comply with all the procedures included in the protocol.

Exclusion Criteria:

Healthy volunteers:

* pregnancy
* breastfeeding
* chronic drug treatment
* non healthy

Waiting List Patients:

* Patients with previous transplant.
* Patients with more of one transplanted organ.
* Patients on anticalcineurin drugs.
* Patients with impaired renal function - creatinine clearance ≤ 20 ml/min.

Transplant Patients:

* Pregnant or breastfeeding.
* Patients with prior retransplantation.
* Patients with more of one transplanted organ.
* Patients with impaired renal function - creatinine clearance ≤ 20 ml/min.
* Everolimus indication at any time during treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers Patients of the Waiting List for Liver Transplantation Liver Transplant recipients on Tacrolimus Liver Transplant Recipients on Cyclosporine Longitudinal Cohort of Patients since their pretransplant condition up 1 year posttransplantation
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of expression of CD25High in CD3, CD4 and CD8 T Lymphocytes. | All subjects at the inclusion. Patients from the longitudinal cohort: at 0, 30, 90, 180 and 360 days post transplantation.
  Related to T lymphocyte activation
Pharmacogenetic investigations | At the moment of the inclusion for all cohorts.
  Related to the influence of genetic variants in anticalcineurin drug pharmacodynamics
Anticalcineurin drug concentration through levels | At the moment of the inclusion and at each regular office visit during check up.
  Related to whole blood target calcineurin inhibitor concentration values
Change in Mean Fluorescence Intensity of NFAT1 Nuclear Translocation Inhibition in PMBC nuclei. | All subjects at the inclusion. Patients from the longitudinal cohort: at 0, 30, 90, 180 and 360 days post transplantation.
  Related to calcineruin activation/inhibition (enzyme target of this group of drugs).
Change in the Percentage of expression of IL-2 in CD4 and CD8 subsets of T lymphocytes. | All subjects at the inclusion. Patients from the longitudinal cohort: at 0, 30, 90, 180 and 360 days post transplantation.
  Related to T cell function and the maintenance of T cell response.

SECONDARY OUTCOMES:
Acute Cellular Rejection Mild, Moderate and Severe | Within the year of follow up.
  Recipients's Immune response to his graft
Infection Episodes which requiere anmicrobials treament | Within the year of follow up
Neurotoxicity to CNIs | Within the year of follow up
Nephrotoxicity to CNIs | Within the year of follow up
Malignancies | Within the year of follow up
Post transplant Diabetes | Within the year of follow up
Cardiovascular disease, post transplant blood pressure augmentation | Within the year of follow up
Death | Within the year of follow up
Post transplant surgical complications | Within the year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ofelia M Noceti, PhD, PharmD, Principal Investigator — National Center for Liver Transplantation and Liver Diseases Department, Hospital Central de las Fuerzas Armadas; Solange Gerona, MD, Study Chair — National Center for Liver Transplantation and Liver Diseases Department, Hospital Central de las Fuerzas Armadas
Locations (1):
- National Center for Liver Transplantation and Liver Diseases Department, Hospital Central de las Fuerzas Armadas, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
Through scientific publications and congresses
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once the trial concludes
Access Criteria: On request

REFERENCES:
- [Derived] Noceti O, Pouche L, Esperon P, Lens D, Vital M, Tourino C, Gerona S, Woillard JB, Marquet P. Activity of the Calcineurin Pathway in Patients on the Liver Transplantation Waiting List: Factors of Variability and Response to Tacrolimus Inhibition. Clin Chem. 2017 Nov;63(11):1734-1744. doi: 10.1373/clinchem.2017.272534. PMID 29054923
- Available data/document: Clinical Study Report: PMID: 25142246 — http://www.ncbi.nlm.nih.gov/pubmed/25142246 — Tacrolimus pharmacodynamics and pharmacogenetics along the calcineurin pathway in human lymphocytes.
- Available data/document: Clinical Study Report: PMID: 29054923 — https://www.ncbi.nlm.nih.gov/pubmed/29054923 — Activity of the Calcineurin Pathway in Patients on the Liver Transplantation Waiting List: Factors of Variability and Response to Tacrolimus Inhibition.